CLINICAL TRIAL: NCT05060302
Title: Prognosis of Right Ventricular Dysfunction Assessed by Speckle Tracking in Postoperative Thoracic Surgery: a Pilot Study
Brief Title: Prognosis of Right Ventricular Dysfunction Assessed by Speckle Tracking in Postoperative Thoracic Surgery
Acronym: SPECKLETHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2021_843_0030
Record Dates: First submitted 2021-09-15; First posted 2021-09-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Right Ventricle; Thoracic Surgery
Keywords: Right ventricle; speckle tracking; thoracic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: transthoracic echocardiography (TTE) — the included patients have a TTE preoperatively in order to evaluate the RV systolic function. TTE will also be done at day 2 and day-15 during the follow-up surgical consultation.

SUMMARY:
In postoperative thoracic surgery (lobe resection, pneumonectomy or wedge resection), cardiovascular complications are the most frequent (10 to 15%) with a significant morbi-mortality rate. Right ventricular (RV) dysfunction is a complication that can be multifactorial in post thoracic surgery. The RV longitudinal shortening fraction (RV-LSF) is a new 2D-STE parameters able to more accurately detect patients with RV dysfunction compared to conventional echocardiographic parameters.

This project is a single-center, prospective, interventional study of patients hospitalized at the Amiens University Hospital for scheduled thoracic surgery. TTE is performed preoperatively, at day 2 and day 15 following the thoracic surgery. Echocardiographic parameters will be measured by an echocardiographic expert in offline with a dedicated software. MACE criteria will be collected at day 2, day 15 and day-30 following the thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years)
* Patient hospitalized at the Amiens University Hospital for scheduled thoracic surgery (lobectomy, pneumonectomy, wedge resection).
* Surgery by thoracotomy or video-assisted thoracic surgery
* Information of the patient and collection of his non-opposition

Exclusion Criteria:

* Patient with poor echogenicity on TTE not allowing evaluation of 2D-STE or conventional parameters of the RV.
* Patient with a rapid supraventricular rhythm disorder (HR > 100) at the time of TTE
* Patient under mechanical ventilation
* Patient under extracorporeal membrane oxygenation
* Patients under guardianship or legal protection
* Patients whose clinical condition does not allow for their non-opposition
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
occurrence of a major cardiovascular event (MACE) | day 30
  MACE is a composite criteria. MACES criteria is defined as the occurrence of at least one of the following events: A cardiovascular death or a documented supraventricular tachycardia (atrial fibrillation and/or flutter) of duration > 30 seconds or, an acute myocardial infarction or, an hospitalization for a right ventricular failure or, an hospitalization for a left ventricular failure.

SECONDARY OUTCOMES:
Variation of RV systolic function from baseline in patients with MACE | at day 1
Variation of RV systolic function from baseline in patients without MACE | at day 1
Variation of RV systolic function from baseline in patients with MACE | at day 2
Variation of RV systolic function from baseline in patients without MACE | at day 2
Variation of RV systolic function from baseline in patients with MACE | at day 15
Variation of RV systolic function from baseline in patients without MACE | at day 15
Variation of RV systolic function from baseline in patients with MACE | within day 30
Variation of RV systolic function from baseline in patients without MACE | within day 30
Assessment of RV systolic function preoperatively | at day 30
occurrence of a postoperative complication | at day 30

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No